CLINICAL TRIAL: NCT07078175
Title: Effectiveness of Xingnao Kaiqiao Acupuncture Compared to Electroacupuncture in Improving Upper Limb Function in Early Stroke Rehabilitation: A Randomized Controlled Trial
Brief Title: Xingnao Kaiqiao Acupuncture vs Electroacupuncture for Post-Stroke Upper Limb Recovery
Acronym: XNKQ-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Nguyen Ngo Le Minh Anh MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr Nguyen Ngo Le Minh Anh MD, PhD, Lecturer, MD, PhD- Faculty of Traditional Medicine, University of Medicine and Pharmacy at Ho Chi Minh City, University of Science Ho Chi Minh City
Organization: University of Science Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XNKQ-StrokeRCT2025
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-01

CONDITIONS: Post-stroke
Keywords: acupuncture; Xingnao Kaiqiao; Stroke Rehabilitation; Motor Recovery; Traditional Medicine
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Participants were randomized in a 1:1 ratio to receive either Xingnao Kaiqiao acupuncture or standard electroacupuncture for 4 weeks. Treatment assignments were parallel with no crossover
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to the treatment allocation to minimize assessment bias. Neither participants nor care providers were masked due to the nature of acupuncture interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xingnao Kaiqiao Acupuncture (Experimental): Participants in this group received Xingnao Kaiqiao (XNKQ) acupuncture based on the standardized protocol developed by Prof. Shi Xuemin, focusing on awakening the brain and opening the sensory orifices. Treatment was administered once daily for 5 days/week over 4 weeks.
  Interventions: Procedure: Xingnao Kaiqiao Acupuncture
- Electroacupuncture (Active Comparator): Participants in this group received routine electroacupuncture therapy applied to standard upper-limb motor recovery acupoints. Treatment was administered once daily for 5 days/week over 4 weeks.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Xingnao Kaiqiao Acupuncture — Acupuncture procedure developed by Prof. Shi Xuemin. Key acupoints include DU26, PC6, SP6, LI4, and GV20, applied with rapid and penetrating stimulation.
  Arm(s): Xingnao Kaiqiao Acupuncture
  Arms: Xingnao Kaiqiao Acupuncture
Procedure: Electroacupuncture — Routine electroacupuncture using standard acupoints for hemiplegic upper limb rehabilitation, including LI15, LI11, SJ5, and LI4, with low-frequency electrical stimulation.
  Arms: Electroacupuncture

SUMMARY:
This is a single-center interventional study conducted at the Ho Chi Minh City Hospital for Orthopedics and Rehabilitation, led by investigators from the University of Medicine and Pharmacy at Ho Chi Minh City. The study aims to evaluate the effectiveness of a specific acupuncture protocol (Xingnao Kaiqiao - Brain Awakening Acupuncture) in improving upper limb motor recovery in post-ischemic stroke patients during the early rehabilitation phase.

Data collection has been completed, and the study is currently being registered on ClinicalTrials.gov to ensure research transparency, ethical compliance, and to facilitate future publication. The final results and publication will be updated once the study receives a registration number.

DETAILED DESCRIPTION:
This single-center interventional study was conducted at the Ho Chi Minh City Hospital for Orthopedics and Rehabilitation under the leadership of investigators from the University of Medicine and Pharmacy at Ho Chi Minh City. The objective of the study was to evaluate the effectiveness of the Xingnao Kaiqiao (Brain Awakening) acupuncture protocol in improving upper limb motor recovery in patients during the early rehabilitation phase following an ischemic stroke.

Eligible participants were screened and recruited according to predefined inclusion and exclusion criteria. Patients received standardized rehabilitation care, and the intervention group additionally received Xingnao Kaiqiao acupuncture targeting key acupoints associated with brain function and motor control. Outcomes were assessed using validated clinical scales and objective motor function tests.

The study adhered strictly to ethical guidelines and was approved by the Biomedical Research Ethics Committee of the University of Medicine and Pharmacy at Ho Chi Minh City (Approval No. 3332/HDDD-DHYD, dated November 6, 2024). Data collection and intervention have been completed, and the results are being prepared for formal analysis and publication. This registration serves to ensure research transparency and compliance with international standards for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 to 80 years
* Diagnosed with ischemic or hemorrhagic stroke confirmed by CT or MRI
* Stroke onset between 1 and 6 months prior to enrollment
* Moderate to severe upper limb motor impairment (FMA-UE score between 20 and 60)
* Medically stable and able to attend treatment sessions 3 times per week
* Capable of understanding the study procedures and providing informed consent

Exclusion Criteria:

* History of severe cognitive impairment (MMSE score < 20)
* Comorbidities that affect motor function (e.g., Parkinson's disease, multiple sclerosis)
* Severe aphasia or communication disorder that prevents assessment
* Botulinum toxin injection in the upper limb within the past 3 months
* Pacemaker or other contraindications to electroacupuncture
* Currently participating in another clinical trial
* Skin infections or local conditions at acupuncture sites

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment of Upper Extremity (FMA-UE) Score | 4 weeks
  Change in FMA-UE score from baseline to 4 weeks post-treatment. The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) is a validated scale that measures upper limb motor function in post-stroke patients.
  The scale ranges from 0 (severe impairment) to 66 (normal function). Higher scores indicate better recovery of motor function.

SECONDARY OUTCOMES:
Change in Barthel Index Score | 4 weeks
  Change in Barthel Index score from baseline to 4 weeks post-treatment to assess improvement in activities of daily living (ADL). The Barthel Index ranges from 0 (completely dependent) to 100 (fully independent). Higher scores indicate better functional independence
Proportion of Participants Achieving MCID in FMA-UE | 4 weeks
  Percentage of participants showing a clinically meaningful improvement in upper extremity motor function, defined as a ≥5-point increase in FMA-UE score from baseline to 4 weeks. This threshold is based on established Minimal Clinically Important Difference (MCID) criteria for post-stroke populations.
Proportion of Participants Achieving MCID in Barthel Index | 4 weeks
  Percentage of participants demonstrating a clinically important improvement in daily functional independence, defined as a ≥10-point increase in Barthel Index score from baseline to 4 weeks. This is considered a meaningful change in functional recovery after stroke.

OTHER OUTCOMES:
Incidence and Classification of Adverse Events | 4 weeks
  The frequency, type, severity, and relationship to treatment of all adverse events (AEs) occurring during the 4-week intervention period. Adverse events include local reactions (e.g., pain, bruising, bleeding), systemic symptoms (e.g., dizziness, fatigue), and serious adverse events (SAEs) as per ICH-GCP criteria. Events will be assessed and documented by blinded evaluators using a standardized adverse event reporting form.
Patient Global Impression of Change (PGIC) | 4 weeks
  Patient self-reported global impression of overall improvement, rated using a 7-point Likert scale ranging from "Very much worse" to "Very much improved," collected at the end of the 4-week treatment period. This scale reflects the patient's perception of treatment benefit and subjective functional change.

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Anh Nguyen Ngo Le, M.D., Ph.D., Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City, Viet Nam
Locations (1):
- Ho Chi Minh City Orthopedic and Rehabilitation Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam